CLINICAL TRIAL: NCT02181465
Title: Phase II, Open Label, Single Center, Two Arm Study Study to Assess the Safety, Tolerance and Efficacy of a 2 mg Dose of G17DT Via Intramuscular Injection in Patients With Advanced Metastatic Colorectal Adenocarcinoma.
Brief Title: Study to Assess Safety and Tolerability of G17DT in Patients With Colorectal Adenocarcinoma.
Acronym: CC1A&B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC1A&B
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

ARMS (2):
- Group 1 (Experimental): One injection of G17DT followed by up to three booster injections depending on antibody response over 16 week period
  Interventions: Biological: G17DT
- Group 2 (Experimental): Three injections of G17DT with option of one booster after 16 weeks
  Interventions: Biological: G17DT

INTERVENTIONS:
Biological: G17DT

SUMMARY:
Pancreatic, gastric, and colorectal cancers have all been shown to overexpress the gastrin gene and to be sensitive to the trophic effects of the gastrin in animal models. The hypothesis of this study is that G17DT will elicit specific and high-affinity antibodies that will bind gastrin-17, thus preventing the trophic activity of cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma of the colon or rectum
* Recurrent/ metastatic disease not amenable to curative surgery and/or radiotherapy
* measurable/ evaluable lesions
* Life expectancy > 3 months
* Karnofsky index > 50% or WHO performance rating of 0-2
* Biochemical markers:

  * renal function < 25% above upper limit of normal range (creatinine, 140 imol/1 unless malignant involvement proven)
  * liver function < 25% above upper limit of normal range (bilirubin ~25 mcmol/1 unless malignant involvement proven)
* Haematological status:

  * haemoglobin, 11 g/ dl
  * WBC, 4 X 109/1
  * platelets, 100 x 109/l
* Written consent

Exclusion Criteria:

* Other concomitant malignant disease except treated basal cell carcinoma of the skin or cancer of the uterine cervix stage 0-1
* H 2 receptor antagonist or proton pump inhibitor therapy
* Previous gastric surgery (including vagotomy)
* Active uncontrolled infection
* Autoimmune disorders
* Anticancer treatment within the last three months unless progression of the disease occurred in the interim
* Women of child-bearing age
* Patient is a poor medical risk because of non-malignant systemic disease
* Previous radiotherapy to all measurable or evaluable lesions.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1993-10; Primary Completion 1994-05 (Actual); Study Completion 1994-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse effects | Up to week 16

SECONDARY OUTCOMES:
Measure serum anti gastrin-17 antibodies to determine immunological response to medication | Up to week 16

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom